CLINICAL TRIAL: NCT03074799
Title: Nurse-Led, Symptom-Based Screening of Household Child Contacts of Tuberculosis Index Cases
Acronym: SOAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00055079
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: We propose a cluster randomized trial to be conducted in 16 decentralized care clinics with existing TB services that will measure the implementation of symptom-based, nurse-led initiation of IPT compared to the current standard of care with TST-based referral to a pediatricians at the district hospital. A baseline assessment of clinic records and procedures will inform clinic stratification prior to randomization. Clinics will be stratified by size (number of patients seen per month) and TB case notifications. The clinics will then be randomized in a 1:1 ratio to receive either the intervention or the current standard of care. Given the intervention will be carried out by a clinic in its entirety, neither the provider nor the patient will be blinded to the study procedure. No additional staff will be provided to the clinics to assist in this process as we wish to evaluate the implementation of IPT for child contacts under 5 years old in a real world, resource-limited setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TST-based Screening (Child contacts) (Active Comparator): In the control clinics, decision regarding IPT will be made based on TST results, as is now the standard of care in this South African health district. In this setting, all TST negative children are initiated on IPT by the nurse at the local clinic. TST positive children are all referred to the district hospital for further evaluation of TB disease regardless of clinical symptoms. Again, clinical outcome data will be obtained from patient records and the same longitudinal child contact register.
  Interventions: Other: Symptom -based Screening(Child Contacts)
- Symptom -based Screening(Child Contacts) (Experimental): In the intervention clinics, decisions regarding IPT will be made on a clinical basis. If the child is symptomatic, they will be referred to the hospital for further evaluation of TB disease including both chest X-ray and testing of either sputum or swallowed sputum. If the child is asymptomatic, the TB nurse at the local clinic will initiate them on weight-appropriate dosing of IPT. Children will be followed at least monthly for the duration of the six month course of isoniazid, as is standard of care in South Africa at this time. Clinical outcome data will be obtained from patient records and implementation of a contact register aimed at improving longitudinal care of children on isoniazid preventive therapy.
  Interventions: Other: Clinical based Decisions

INTERVENTIONS:
Other: Symptom -based Screening(Child Contacts) — Aim 1: Determine the number of child contacts per adult index case of tuberculosis to assess quality of contact tracing.
  Aim 2: Determine the percentage of child contacts initiated on IPT or antituberculous therapy (ATT) and compare between intervention (symptom-based, nurse-led initiation of IPT) vs control clinics (TST-based screening with referral to hospital, current standard of care).
  Aim 3: Compare outcomes of children initiated on IPT between both groups including: completion of therapy, discontinuation due to side effects, lost to follow up, and adherence while on therapy.
  Arms: TST-based Screening (Child contacts)
Other: Clinical based Decisions — the child is symptomatic, they will be referred to the hospital for further evaluation of TB disease including both chest X-ray and testing of either sputum or swallowed sputum. If the child is asymptomatic, the TB nurse at the local clinic will initiate them on weight-appropriate dosing of IPT
  Arms: Symptom -based Screening(Child Contacts)

SUMMARY:
To assess implementation of a nurse-led, symptom-based screening program in local, decentralized clinics for tuberculosis (TB) screening of child contacts less than 5 years old who were exposed to tuberculosis in the home. This will allow nurses in decentralized clinics to either start IPT for those asymptomatic patients and refer symptomatic patients for evaluation of TB disease and possible antituberculous therapy (ATT).

DETAILED DESCRIPTION:
Retrospective review of routine program data for child contacts less than five years of adult TB index cases who are receiving TB care at local, decentralized clinics in the Matlosana district of Northwest Province will be assessed. 16 clinics will be stratified and randomized in 1:1 fashion to either TST-based screening, the current standard of care, or symptom-based screening, the newly recommended standard of care in South Africa. Those who are TST positive in the TST-based group and those who are symptomatic in the symptom-based group will be referred to Klerkdorp Hospital for further evaluation of tuberculosis. Nurses in the decentralized clinics will initiate those who are TST negative or asymptomatic on IPT. Their clinical course will be monitored throughout treatment and adherence to therapy measured. The investigators will compare clinic-level outcomes including percentage of patients initiated on, adherent to, and completing IPT.

ELIGIBILITY:
Inclusion Criteria:

* Child less than five years old
* Household contact of a drug-sensitive pulmonary or extrapulmonary TB index case (drug sensitivity is define as culture-confirmed OR absence of rifampin resistance on gene Xpert) admitted to one of the public clinics in the Matlosana sub-district on or after October 1, 2015.

Exclusion Criteria:

* Household contact of a drug-resistant TB index case. (Drug resistance defined either by culture or by presence of rifampin resistance on gene Xpert).

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4054 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Percent of child contacts placed on IPT | 2 years
  The primary outcome is the mean percentage of identified contacts initiated on IPT or ATT

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chaisson, MD, Principal Investigator — Director, Center for Tuberculosis Research
Locations (1):
- PHRU, Klerksdorp, Matlosana, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Study is ongoing; plans for data sharing are in process

REFERENCES:
- [Derived] Salazar-Austin N, Milovanovic M, West NS, Tladi M, Barnes GL, Variava E, Martinson N, Chaisson RE, Kerrigan D. Post-trial perceptions of a symptom-based TB screening intervention in South Africa: implementation insights and future directions for TB preventive healthcare services. BMC Nurs. 2021 Feb 8;20(1):29. doi: 10.1186/s12912-021-00544-z. PMID 33557831
- [Derived] Salazar-Austin N, Cohn S, Barnes GL, Tladi M, Motlhaoleng K, Swanepoel C, Motala Z, Variava E, Martinson N, Chaisson RE. Improving Tuberculosis Preventive Therapy Uptake: A Cluster-randomized Trial of Symptom-based Versus Tuberculin Skin Test-based Screening of Household Tuberculosis Contacts Less Than 5 Years of Age. Clin Infect Dis. 2020 Apr 10;70(8):1725-1732. doi: 10.1093/cid/ciz436. PMID 31127284